CLINICAL TRIAL: NCT04497168
Title: Citalopram as a Posterior Cortical Protective Therapy in Parkinson Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Vikas Kotagal, Associate Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00146905; 1R01AG065246 (NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Serotonin; Selective Serotonin Reuptake Inhibitor; Amyloid-beta
MeSH Terms: conditions — Parkinson Disease; Plaque, Amyloid | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Citalopram (Experimental): 20mg daily
  Interventions: Drug: Citalopram 20mg
- Placebo (Placebo Comparator): matching placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram 20mg — 20mg daily
  Arms: Citalopram
Drug: Placebo — matching placebo pills
  Arms: Placebo

SUMMARY:
This Parkinson disease (PD) trial will test whether 26 months of citalopram, compared to placebo, can alter the build-up of toxic amyloid-beta plaques in the visuospatial cortex of the brain linked to visuospatial cognitive impairment in PD.

DETAILED DESCRIPTION:
This study is a proof-of-concept Parkinson disease trial aimed at delaying visuospatial cognitive decline, an important component of Parkinson dementia. In Parkinson disease, low-range cortical Abeta plaque levels associate with serotonin terminal losses. Multicenter Parkinson disease observational findings show that selective serotonin reuptake inhibitors (SSRIs) associate with lower dementia conversion risk and different cerebrospinal fluid Abeta-42 levels. This study aims to test the hypothesis that citalopram use in Parkinson disease will reduce visuospatial cortex Abeta plaque accrual, leading to an amelioration of longitudinal visuospatial cognitive decline linked to Parkinsonian dementia. The study will test this hypothesis in a randomized placebo-controlled trial of citalopram 20mg daily over 26 months in Parkinson disease subjects (age ≥65) without depression (n=58).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a Parkinson Disease (PD) diagnosis based on the United Kingdom Parkinson's Disease Society Brain Bank Research Center clinical diagnostic criteria
* Modified Hoehn and Yahr (HY) scores spanning 2.0 to 3.0
* Age 65 years or greater

Exclusion Criteria:

* Diagnosis of an atypical parkinsonian condition
* Participants on neuroleptics and participants with a history of use of anti-depressants (including selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), bupropion, St. John's Wort or other serotoninergic agents in the year preceding study enrollment
* Evidence of a large artery stroke or mass lesion on brain imaging
* Participants with a life threatening comorbid illness
* Severe claustrophobia precluding PET imaging
* Inability to participate in research procedures involving ionizing radiation
* Pregnancy or breastfeeding
* Participants with active depression as defined by a Geriatric Depression Scale score of >10 or on the basis of clinical diagnosis by the PI
* Participants who report active suicidal ideation as defined by an affirmative answer to questions 1 and 2 on the C-SSRS
* Participants with baseline HY scores <2.0 or ≥3.0
* Participants with a QTc interval on baseline EKG >0.45 for men or >0.47 for women
* Subjects taking certain contraindicated medications at baseline
* Subjects unable to swallow pills
* Subjects with a previous history of mania, ongoing hepatic impairment or epilepsy
* Subjects with a known allergy to citalopram or escitalopram
* Subjects with substantial cognitive impairment or dementia that would prevent them from providing informed consent
* Subjects in another ongoing clinical trial
* Subjects with treatment-naieve Parkinson disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in visuospatial cortex PiB distribution volume ratio (DVR) | Baseline to month 26
  PiB PET can assess the density of amyloid-beta plaques in the brain. This imaging method will be used to quantify the amount of change in amyloid-beta plaques levels--measured specifically within the visuospatial cortex--between month 0 and month 26.

SECONDARY OUTCOMES:
Change in Benton Judgement of Line Orientation (JOLO) test score | Baseline to month 26
  This is a standardized test with 30 items that is specific for visual spatial cognition. The minimum score is 0, indicating low visual spatial cognition. The maximum score is 30, indicating high visual spatial cognition.
Change in Montreal Cognitive Assessment (MoCA) score | Baseline to month 26
  This scale evaluates different domains of cognition like attention, orientation, memory, language, visuoconstructional capacities, and lastly, executive functions. MoCA is a 30 point test with lower scores indicating impaired cognition. The maximum score is 30.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Kotagal, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be uploaded in a timely manner in the "openICPSR" Data Management Resource (DMR) of ICPSR (Inter-University Consortium for Political and Social Research). Biospecimens (DNA) will be banked in the NIA NCRAD biorepository. Uploaded datasets will be stripped of identifiers in order to prevent the possibility of identifying human subjects participants in this study from the publically available dataset.
Supporting Information: Study Protocol
Time Frame: Consistent with NIA policies, the study team will ensure the dataset is shared by the occurrence of the earlier of the following two milestones: either the date of primary publication or within 9 months of lifting of the data lock.
Access Criteria: Access to the coded dataset that is uploaded to openICPSR is available to any individual who applies to the openICPSR for data access. This process involves providing a brief description of the intended use of the data to be downloaded, a data use agreement and data security plan, and documentation of IRB approval or exemption.
URL: https://www.openicpsr.org/openicpsr/